CLINICAL TRIAL: NCT03401203
Title: A Prospective, Open Label, Multi-center, Dual Arm, Randomized Trial : The ROTA-ISR (Debulking With Rotational Atherectomy Versus Balloon Angioplasty In Patients With In-stent Restenosis) Trial
Brief Title: Debulking With Rotational Atherectomy Versus Balloon Angioplasty In Patients With In-stent Restenosis
Acronym: ROTA-ISR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, Professor, Division of Cardiology, Asan Medical Center, University of Ulsan, College of Medicine, Seoul, South Korea, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMCCV2017-11
Record Dates: First submitted 2017-12-25; First posted 2018-01-17 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Coronary Vessels
Keywords: ISR; ROTA; DEB; PCI
MeSH Terms: interventions — Angioplasty, Balloon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rotational atherectomy followed by balloon angioplasty (Experimental)
  Interventions: Procedure: Rotational atherectomy followed by balloon angioplasty
- balloon angioplasty (Active Comparator)
  Interventions: Procedure: Balloon angioplasty

INTERVENTIONS:
Procedure: Rotational atherectomy followed by balloon angioplasty — Percutaneous coronary intervention
  Arms: rotational atherectomy followed by balloon angioplasty
Procedure: Balloon angioplasty — Percutaneous coronary intervention
  Arms: balloon angioplasty

SUMMARY:
This study is to establish the primary hypothesis that debulking with rotational atherectomy (RA) followed by balloon angioplasty (BA) is superior to BA alone for lesion preparation in patients with coronary in-stent restenosis (ISR) regarding angiography-measured in-segment minimal lumen area at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Men or women at least 19 years of age
* Subjects with coronary In-stent restenosis planned revascularization
* In-stent restenosis with neointimal hyperplasia evaluated by intravascular imaging
* The patient or guardian agrees to the study protocol and the schedule of clinical follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site.

Exclusion Criteria:

* Complex lesion anatomy that disables rotational atherectomy
* Any clinically significant abnormality identified at the screening visit, physical examination, laboratory tests, or electrocardiogram which, in the judgment of the Investigator, would preclude safe completion of the study.
* Life expectancy < 1 years for any non-cardiac or cardiac causes
* Unwillingness or inability to comply with the procedures described in this protocol.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
In-segment minimal lumen diameter on angiographic | 1 year

SECONDARY OUTCOMES:
Device success rate | 1 year
Angiographic outcomes immediate after procedure | 1 hour
  In-segment and in-stent minimal lumen diameter and diameter stenosis
OCT outcomes immediate after procedure : In-segment and in-stent minimal lumen area | 1 hour
OCT outcomes immediate after procedure : In-segment and in-stent neointimal volume | 1 hour
Angiographic outcomes : In-segment and in-stent late loss, diameter stenosis | 1 year
OCT outcomes : in-segment and in-stent late lumen area, minimal lumen area loss | 1 year
composite event rate | 1 year
  A composite event of following factors is defined as the occurrence of any event from these events and denoted that event as the union of these.
  * Death (cardiac, vascular, non-cardiovascular)
  * Myocardial infarction (periprocedural, spontaneous)
  * Stent thrombosis (definite/probable)
  * Stroke
  * Any revascularization
  * Target lesion revascularization (TLR)
  * Target vessel revascularization (TVR)
  * Clinically significant bleeding (BARC type 2,3,4,5)
  * Target lesion failure (cardiac death, target vessel MI or ischemia-driven TLR)
  * Target vessel failure (cardiac death, target vessel MI or ischemia-driven TVR)
  * A composite of all-cause death, MI, any repeat revascularization
  * A composite of cardiac death, target vessel MI, stroke, or clinically significant bleeding (Bleeding Academic Research Consortium (BARC) type 2,3,4,5)

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - Chonnam National University Hospital, Gwangju
  - Asan Medical Center, Seoul